CLINICAL TRIAL: NCT07241507
Title: Frequency of Wound Dehiscence and Wound Infection in Continuous Versus Interrupted Suturing for Abdominal Closure in Exploratory Laparotomy
Brief Title: Effect of Continuous Versus Interrupted Suturing on Wound Dehiscence and Infection After Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Shehroz Sarwar, Principal Investigator, Allama Iqbal Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1329-8430
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Laparotomy Closure After Abdominal Surgery; Wound Infection, Surgical; Dehiscence of Laparotomy Wound; Suture, Interrupted; Continuous Suture
Keywords: exploratory laparotomy; Surgical wound infection; Wound dehiscence
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Continuous (Active Comparator): Continuous Suture
  Interventions: Procedure: Continuous suturing
- Group B - Interrupted (Experimental): Interrupted Suture
  Interventions: Procedure: Interrupted suturing

INTERVENTIONS:
Procedure: Continuous suturing — After an exploratory laparotomy continuous suturing using a single thread of Vicryl No. 1 will be used to stitch the incision's fascial layer together, 1 cm distance from wound edges and between each stitch, creating a line of even tension across the wound.
  Arms: Group A - Continuous
Procedure: Interrupted suturing — After an exploratory laparotomy, interrupted suturing using a single thread of Vicryl No. 1 will be used to stitch the incision's fascial layer together, 1 cm distance from wound edges and between each stitch. A knot will be tied after each suture is passed through the tissue, and each stitch will be secured with its own knot.
  Arms: Group B - Interrupted

SUMMARY:
The goal of this clinical trial is to learn whether the type of suturing technique used to close the abdomen after exploratory laparotomy affects the rate of wound complications. Specifically, the study aims to find out if using interrupted sutures results in fewer cases of wound dehiscence (wound reopening) compared to continuous sutures.

The main question the study seeks to answer is:

Does interrupted suturing reduce the frequency of wound dehiscence compared to continuous suturing in patients undergoing exploratory laparotomy?

Researchers will also observe and compare wound infection rates between the two suturing methods.

About 80 adult patients (18-60 years old) undergoing exploratory laparotomy at the Department of General Surgery, DHQ Teaching Hospital, Dera Ghazi Khan, will take part in this study. Participants will be randomly assigned to one of two groups:

Group A: Continuous abdominal closure using No. 1 Vicryl suture

Group B: Interrupted abdominal closure using No. 1 Vicryl suture

All participants will have their baseline characteristics recorded, including age, gender, obesity, diabetes, and smoking status. The surgical technique and postoperative care will follow the hospital's standard protocols. After surgery, patients will be followed for four weeks with weekly clinical assessments to check for wound infection or wound dehiscence.

The hypothesis is that patients whose abdominal wounds are closed with interrupted sutures will have a lower frequency of wound dehiscence compared to those with continuous sutures.

The findings will help guide surgeons on which abdominal closure method provides better wound healing and fewer postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing exploratory laparotomy
* Both emergency and elective

Exclusion Criteria:

* Patients undergoing second laparotomy or re- laparotomy
* Patients on steroid therapy (assessed on medical record review)
* Patients who die within 28-days of surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Wound Dehiscence | From enrollment to 28-days of operation
  A partial or total separation of previously approximated wound edges, on clinical examination of surgical wound.

OTHER OUTCOMES:
Surgical Wound Infection | From enrollment to 28-days after operation
  Presence any features of erythema, pain, pus discharge on examination of surgical wound and new onset fever (> 98.60F)

CONTACTS AND LOCATIONS:
Overall Officials: Malik N Fareed, FCPS, Study Chair — Allama Iqbal Teaching Hospital Dera Ghazi Khan
Locations (1):
- Allama Iqbal Teaching Hospital, Dera Ghazi Khan, Dera Ghazi Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No